CLINICAL TRIAL: NCT06189586
Title: Comparison of Aerosol Inhalation and Intravenous Glucocorticoid in the Treatment of Severe AECOPD-------Multicenter, Prospective, Randomized, Controlled Clinical Study
Brief Title: Comparison of Aerosol Inhalation and Intravenous Glucocorticoid in the Treatment of Severe AECOPD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Dong Yang (Other)
Collaborators: Jilin University (Other)
Responsible Party: Sponsor-Investigator, Dong Yang, Assisted Investigator, Jilin University
Organization: Jilin University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 130064
Record Dates: First submitted 2023-12-19; First posted 2024-01-03 (Actual); Last update posted 2024-01-03 (Actual); Status verified 2023-12

CONDITIONS: Acute Exacerbation of Chronic Obstructive Pulmonary Disease
Keywords: severe AECOPD; aerosol inhalation and intravenous glucocorticoid

STUDY DESIGN:
Intervention Model Description: Description for medicine or protocol of treatment in detail:
  Dosing regimen:
  1. Intravenous hormone group: 40mg sodium methylprednisolone succinate for injection(dissolved in 0.9% saline or5% glucose injection 50ml), intravenous infusion for 30 minutes, once a day for 5 consecutive days.
  2. Nebulized inhalation group: 2 mg budesonide suspension for inhalation, nebulized inhalation for minutes,administered 4 times a day for 5 consecutive days.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nebulized inhalation group (Active Comparator): 2 mg budesonide suspension for inhalation, nebulized inhalation for minutes,administered 4 times a day for 5 consecutive days.
  Interventions: Drug: aerosol inhalation of glucocorticoids
- Intravenous hormone group (Active Comparator): 40mg sodium methylprednisolone succinate for injection(dissolved in 0.9% saline or5% glucose injection 50ml), intravenous infusion for 30 minutes, once a day for 5 consecutive days.
  Interventions: Drug: intravenous injection of glucocorticoids

INTERVENTIONS:
Drug: aerosol inhalation of glucocorticoids — Patients with severe AECOPD were continuously recruited from the care unit of Respiratory and Critical Care Medicine Department of the First Hospital of Jilin University to conduct a randomized cohort study, which was divided into aerosol inhalation group and intravenous glucocorticoid group. Subjects in the intravenous hormone group received 40mg methylprednisolone (dissolved in 0.9% normal saline /5% glucose injection 50ml) intravenously once a day. It lasts for 5 days. The atomized inhalation
  Arms: Nebulized inhalation group
Drug: intravenous injection of glucocorticoids — Patients with severe AECOPD were continuously recruited from the care unit of Respiratory and Critical Care Medicine Department of the First Hospital of Jilin University to conduct a randomized cohort study, which was divided into aerosol inhalation group and intravenous glucocorticoid group. Subjects in the intravenous hormone group received 40mg methylprednisolone (dissolved in 0.9% normal saline /5% glucose injection 50ml) intravenously once a day. It lasts for 5 days. The atomized inhalation
  Arms: Intravenous hormone group

SUMMARY:
Comparison of aerosol inhalation and intravenous glucocorticoid in the treatment of severe AECOPD-------Multicenter, prospective, randomized, controlled clinical study

DETAILED DESCRIPTION:
This study aims to compare the efficacy and comprehensive benefits of aerosol inhalation and intravenous injection of glucocorticoids in severe AECOPD patients.

ELIGIBILITY:
Inclusion Criteria:

(1) Patients with AECOPD requiring hospitalization or emergency treatment (COPD acute attacks combined with respiratory failure were eligible). (2) 18 years of age ≤80 years of age (3) Patients and their families are willing to participate in clinical research and sign informed consent.

Exclusion Criteria:

1. Combined with tuberculosis.
2. Combined bronchiectasis.
3. complicated with definite infectious diseases.
4. PCT≥0.5ng/ml or CRP≥30mg/L.
5. Serious injury combined with other organ functions
6. Contraindications to other glucocorticoid use.
7. Concomitant bronchial asthma or positive bronchodilation test

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2021-10-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-07-31 (Estimated)

PRIMARY OUTCOMES:
Relevant indexes after treatment | The day of admission, day one, day two, day three, day five, day seven, day ten
  Changes in blood gas indexes (oxygenation index, arterial partial pressure of carbon dioxide, pH value) of patients with respiratory rate, blood pressure, heart rate changes

CONTACTS AND LOCATIONS:
Overall Officials: Dan Li, Doctor, Study Director — The First Hospital of Jilin University
Locations (1):
- The First Hospital of Jilin University, Changchun, Jilin, China

IPD SHARING:
Plan to Share IPD: No